CLINICAL TRIAL: NCT03941418
Title: Impact of Additional Treatment With Saccharomyces Boulardii on Quality of Life in Patients With Mild Forms of Ulcerative Colitis and Crohn Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Clinic Dr Dragisa Misovic-Dedinje (Other)
Collaborators: University Clinic Zvezdara (Unknown)
Responsible Party: Principal Investigator, Nikola Panic, MD, PhD, University Clinic Dr Dragisa Misovic-Dedinje
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCDragisaMisovic1
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis; Crohn Disease
Keywords: Saccharomyces boulardii
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boulardii (Experimental): Patients will be administered with formulation containing 500 mg of Saccharomyces boulardii and 10 mg of Vitamin D3 once daily, as an addition to their standard therapy.
  Interventions: Dietary Supplement: Boulardii
- Placebo (Placebo Comparator): Patients will be administered with placebo as an addition to their standard therapy.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Boulardii — Patients will be administered with formulation containing 500 mg of Saccharomyces boulardii and 10 mg of Vitamin D3 once daily, as an addition to their standard therapy.
  Arms: Boulardii
Dietary Supplement: Placebo — Patients will be administered with placebo of same appearance, colour and taste once daily.
  Arms: Placebo

SUMMARY:
The goal of the study is to assess the impact of treatment with dietary supplement containing Saccharomyces boulardii (used as an addition to standard therapy), on quality of life of patients with mild forms of ulcerative colitis and Crohn disease, as well as those in remission fulfilling criteria for irritable bowel syndrome.

Patients included will be randomly assigned in two groups and subsequently administered with formulation containing Saccharomyces boulardii or placebo for 4 weeks. Patient's quality of life will be assessed by questionnaire at the enrolment and 4 weeks after initiating the therapy.

DETAILED DESCRIPTION:
Saccharomyces boulardii has been reported to have positive impact on intestinal epithelial barrier as well as immune system. It has been proven to be efficient in treatment and prophylaxis of travellers diarrhoea, HIV associated diarrhoea, antibiotics associated diarrhoea and Clostridium difficile infection. However there is a limited data available on effect of therapy with Saccharomyces boulardii (as add-on to standard therapy) in patients with inflammatory bowel disease. Nevertheless, knowing the effect Saccharomyces boulardii has on intestinal flora, intestinal epithelium and immune system it can be hypothesised that Saccharomyces boulardii used as add-on to standard therapy in IBD patients can lead to improvement in symptoms and therefore in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of ulcerative colitis or Crohn disease
* colonoscopy in last six months confirming mild disease form according to endoscopic criteria (Mayo score, simple endoscopic score)
* colonoscopy in last six months confirming endoscopic remission with fulfilled clinical Rome IV criteria for irritable bowl syndrome
* patients
* patients with mild disease form are eligible only if treated with mesalazine only
* patients in remission eligible for inclusion if treated with mesalazine, biologics, azathioprine or methotrexate
* signed informed consents

Exclusion Criteria:

* no colonoscopy in last six months
* moderate to severe disease according to colonosopy findings (Mayo score, simple endoscopic score)
* indeterminate colitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Patients quality of life | 8 weeks
  Quality of life measured will be measured by questionnaire at day 1, 4 weeks after enrolment and 8 weeks after enrolment.
  Questionnaire comprises 10 questions considering presence of symptoms of inflammatory bowel disease as well as their effect on well-being. Each question can be answered with one of seven answers contributing 1 to 7 points to final score. Final score ranges between 10 and 70 with higher values corresponding with higher quality of life.

SECONDARY OUTCOMES:
Disease clinical activity | 8 weeks
  Disease clinical activity will be measured by Mayo score for ulcerative colitis and Harvey-Bardshaw index for Crohn disease at day 1, 4 weeks after enrolment and 8 weeks after enrollment. The Mayo Score evaluates ulcerative colitis activity based on four clinical parameters. Each parameter of the Mayo score ranges from zero (normal or inactive disease) to 3 (severe activity). The Harvey-Bradshaw index for assessing clinical activity in patients with Crohn disease consists of 5 clinical parameters. Calculation formula for both scores considered the sum of the scores of all the parameters included. Higher values of the score are associated with increased clinical activity of the disease.

IPD SHARING:
Plan to Share IPD: No